CLINICAL TRIAL: NCT01641744
Title: Birth to Three: A Pragmatic Clinical Trial for Child Maltreatment Prevention
Brief Title: Efficacy of Group Attachment Based Intervention for Vulnerable Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: The New School (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Bonuck, Karen A. Bonuck, PhD (Professor), Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-703
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Child Maltreatment; Domestic Violence
Keywords: Parent Child Relationship; Maltreatment; Risk Behaviors; Social and Emotional Development; Violence and Abuse; Policy
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Attachment Based Intervention (GABI) (Experimental)
  Interventions: Behavioral: Group Attachment Based Intervention (GABI)
- Systematic Training for Effective Parenting (STEP) (Active Comparator)
  Interventions: Behavioral: Systematic Training for Effective Parenting (STEP)

INTERVENTIONS:
Behavioral: Systematic Training for Effective Parenting (STEP) — Parenting skills training class, 1x/week, 12 weeks
  Arms: Systematic Training for Effective Parenting (STEP)
Behavioral: Group Attachment Based Intervention (GABI) — Parent-child group, 3x/week, 26 weeks
  Arms: Group Attachment Based Intervention (GABI)

SUMMARY:
The study examines the effectiveness of parent-child Group Attachment Based Intervention (GABI) in reducing risk of maltreatment in infants and toddlers compared with parenting skills classes. GABI directly addresses the needs of isolated, marginalized families, with the goals of of enhancing parent coping and resilience, and improving parent-child attachment relationships.

We hypothesize that compared to usual care, GABI will be associated with improved child, parent and parent-child outcomes.

DETAILED DESCRIPTION:
Child abuse and neglect ("maltreatment") pose enormous short- and long-term risks to children. Yet despite the critical importance of the U.S. Department of Health and Human Services, Maternal and Child Health Bureau's goal "to reduce fatal and non-fatal child maltreatment," non-empirically supported parenting skills classes remain child welfare agencies' standard approach to meeting this goal.

The study examines the effectiveness of parent-child Group Attachment Based Intervention (GABI) in reducing risk of maltreatment in infants and toddlers compared with parenting skills classes. GABI directly addresses the needs of isolated, marginalized families, with the goals of of enhancing parent coping and resilience, and improving parent-child attachment relationships.

Seventy families with children aged 2-36 months who are referred for parenting help will be randomly assigned to either GABI or "treatment as usual" that consists of parents-only parenting skills classes. Treatment will be offered for up to 6 months. Both groups will be assessed at baseline, end of treatment and at 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children age 0-36 months
* Parent(s) is/are biological parent of child (mother or father)
* Parent(s) has/have custody of their child even if he/she/they have lost custody of previous children
* Risk of maltreatment from referral source or intake interview, including parent's own childhood adversity, parent's current exposure to relationship violence, history of parental substance abuse or history of parental incarceration
* If history of substance abuse, enrolled in treatment program
* Willing to sign informed consent

Exclusion Criteria:

* Parent is unable to provide informed consent due to cognitive impairment
* Parent not fluent in English
* Child has diagnosis of an autistic spectrum disorder or severe cognitive delay

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in child exposure to trauma and maltreatment to end-of-treatment and at 6-month follow-up (Child Adverse Childhood Experiences Screener) | Measured at Baseline, End-of-Treatment (12 Weeks for Control/26 Weeks for Intervention), and at 6-Month Follow-up

SECONDARY OUTCOMES:
Child cognitive development (Bayley III Screening Test) | Measured at Baseline, End-of-Treatment (12 Weeks for Control/26 Weeks for Intervention), and at 6-Month Follow-Up
Parent mental health (Symptoms Checklist-90) | Measured at Baseline, End-of-Treatment (12 Weeks for Control/26 Weeks for Intervention), and at 6-Month Follow-Up
Child social-emotional development (Ages and Stages Questionnaire) | Measured at Baseline, End-of-Treatment (12 Weeks for Control/26 Weeks for Intervention), and at 6-Month Follow-Up
Parent social support (Interpersonal Support Evaluation List) | Measured at Baseline, End-of-Treatment (12 Weeks for Control/26 Weeks for Intervention), and at 6-Month Follow-Up
Parenting stress (Parenting Stress Index) | Measured at Baseline, End-of-Treatment (12 Weeks for Control/26 Weeks for Intervention), and at 6-Month Follow-Up
Child-parent attachment (Strange Situation Procedure) and Free -Play Observation coded with Coding Interactive Behavior (CIB) dimensions | Measured at Baseline, End-of-Treatment (12 Weeks for Control/26 Weeks for Intervention, and at 6-Month Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Karen Bonuck, PhD, Principal Investigator — Albert Einstein College of Medicine; Anne Murphy, PhD, Principal Investigator — Albert Einstein College of Medicine; Miriam Steele, PhD, Study Director — The New School; Howard Steele, PhD, Study Director — The New School
Locations (1):
- Center for Babies, Toddlers and Families, division of The Early Childhood Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219